CLINICAL TRIAL: NCT05560464
Title: A Phase 1, Open-label Study to Evaluate the Pharmacokinetics and Safety of Multiple Doses of VX-548 in Subjects With Mild or Moderate Hepatic Impairment and in Matched Healthy Subjects
Brief Title: Evaluation of the Pharmacokinetics and Safety of VX-548 in Participants With Mild or Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VX21-548-007
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Mild Hepatic Impairment (Experimental): Participants will receive multiple doses of VX-548 every 12 hours (q12h) from Day 1 through Day 14.
  Interventions: Drug: VX-548
- Cohort 2: Matched Healthy Participants (Experimental): Healthy participants matched to cohort 1 will receive multiple doses of VX-548 q12h from Day 1 through Day 14.
  Interventions: Drug: VX-548
- Cohort 3: Moderate Hepatic Impairment (Experimental): Participants will receive multiple doses of VX-548 q12h from Day 1 through Day 14.
  Interventions: Drug: VX-548
- Cohort 4: Matched Healthy Participants (Experimental): Healthy participants matched to cohort 3 will receive multiple doses of VX-548 q12h from Day 1 through Day 14.
  Interventions: Drug: VX-548

INTERVENTIONS:
Drug: VX-548 — Tablets for oral administration.
  Other Names: Suzetrigine

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of multiple doses of VX-584 in participants with mild or moderate hepatic impairment as compared to matched healthy controls.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4) (A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Cohorts 1 and 3: Participants with Mild or Moderate Hepatic Impairment

  * Participants will satisfy the criteria for mild (Cohort 1) and moderate hepatic impairment (Cohort 3) defined as a Child-Pugh total score of 5 to 6 and 7 to 9 points, respectively at the screening visit
  * Participants will have chronic (greater than or equal to (≥) 6 months) documented liver disease
* Cohorts 2 and 4: Matched Healthy Participants

  * Participants will be matched (cohort 2 matched to cohort 1; and cohort 4 matched to cohort 3) during screening to participants with hepatic impairment for age, sex, and weight

Key Exclusion Criteria:

* Cohorts 1 and 3: Participants with Mild or Moderate Hepatic Impairment

  * History of febrile illness or other acute illness that has not fully resolved by 14 days before the first dose of study drug
  * Severe portal hypertension
  * History or presence of severe hepatic encephalopathy (Grade >2)
  * Any condition possibly affecting drug absorption
  * Significant renal dysfunction (creatinine clearance <60 milliliter per minute [mL/min] ) estimated according to the method of Cockcroft and Gault at the screening Visit or Day-1
  * History of solid organ or bone marrow transplantation
* Cohorts 2 and 4: Matched Healthy Participants

  * History of febrile illness or other acute illness that has not fully resolved by 14 days before the first dose of study drug
  * Any condition possibly affecting drug absorption

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of VX-548 | Day 1 to Day 31
Area Under the Plasma Concentration Versus Time Curve During a Dosing Interval (AUCtau) of VX-548 | Day 1 to Day 31
Time Taken for VX-548 to Reach Maximum Concentration (tmax) | Day 1 to Day 31
Time Required for Plasma Concentration of VX-548 to Reduce to Half (t1/2) | Day 1 to Day 31
Apparent Volume of Distribution of VX-548 (Vz/F) | Day 1 to Day 31
Apparent Clearance of VX-548 (CL/F) | Day 1 to Day 31
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to the Last Measured Concentration (AUC0-last) of VX-548 | Day 1 to Day 31

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of VX-548 Metabolite | Day 1 to Day 31
Area Under the Plasma Concentration Versus Time Curve During a Dosing Interval (AUCtau) of VX-548 Metabolite | Day 1 to Day 31
Time Taken for VX-548 metabolite to Reach Maximum Concentration (tmax) | Day 1 to Day 31
Time Required for Plasma Concentration of VX-548 Metabolite to Reduce to Half (t1/2) | Day 1 to Day 31
Apparent Volume of Distribution of VX-548 Metabolite (Vz/F) | Day 1 to Day 31
Apparent Clearance of VX-548 Metabolite (CL/F) | Day 1 to Day 31
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to the Last Measured Concentration (AUC0-last) of VX-548 Metabolite | Day 1 to Day 31
Fraction Unbound (fu) for VX-548 and its Metabolite in Plasma | Day 14: Up to 24 hours Post-dose
Unbound Area Under the Concentration Versus Time Curve of VX-548 and its Metabolite | Day 14: Up to 24 hours Post-dose
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 42

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Division of Clinical Pharmacology, University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Oklahoma

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing